CLINICAL TRIAL: NCT00050609
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Study of IC351 (LY450190) in Patients With Diabetic Gastroparesis
Brief Title: Study of Tadalafil for the Treatment of Diabetic Patients With Symptoms of Upset Stomach and Delayed Stomach Emptying
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4979; H6D-MC-LVDC
Record Dates: First submitted 2002-12-16; First posted 2002-12-18 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Active Comparator): 5 mg tadalafil
  Interventions: Drug: tadalafil
- 3 (Active Comparator): 20 mg tadalafil
  Interventions: Drug: tadalafil

INTERVENTIONS:
Drug: tadalafil — 5 mg tadalafil tablet taken by mouth once a day for 8 weeks
  Other Names: LY450190; Cialis; IC351
  Arms: 2
Drug: tadalafil — 20 mg tadalafil tablet taken by mouth once a day for 8 weeks
  Other Names: LY450190; Cialis; IC351
  Arms: 3
Drug: placebo — Placebo tablet taken by mouth once a day for 8 weeks
  Arms: 1

SUMMARY:
The purposes of this study are to determine whether an experimental drug known as tadalafil can reduce symptoms of dyspepsia (fullness after eating, inability to finish a regular meal, bloating, discomfort or pain in the upper abdomen, belching after meals, nausea, vomiting) in diabetic patients, and/or reduce the amount of time the stomach takes to empty the contents of a standard meal. The safety of tadalafil given once daily for 8 weeks in this population will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus
* Delayed gastric emptying
* 3 month minimum history of chronic upper abdominal discomfort
* Symptoms of dyspepsia (upset stomach)

Exclusion Criteria:

* Major gastrointestinal surgery or medical conditions known to affect gastric motility
* Irritable Bowl Syndrome
* Medications known to affect gastric motility
* Angina treated with nitrates
* Uncontrolled diabetes mellitus and history of certain heart problems

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2003-02; Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Measure of change from baseline to endpoint using the Total Symptom Severity Score in patients taking 5 mg tadalafil compared to placebo | 8 weeks

SECONDARY OUTCOMES:
Measure of change from baseline to endpoint using the Total Symptom Severity Score in patients taking 20 mg tadalafil compared to placebo | 8 weeks
Measure of change from baseline to endpoint using the Visual Analog Score and Nepean Dyspepsia Index Symptom Checklist in patients taking 5 mg tadalafil, 20 mg tadalafil and placebo | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- Canada (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmonton, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Victoria, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Courtice, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kitchener, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sainte-Foy, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saskatoon, Saskatchewan

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com